CLINICAL TRIAL: NCT06723002
Title: Effect of Olive Leaf Extracts on Endothelial Dysfunction and Short-term Outcome in Patients With Acute Coronary Syndrome
Brief Title: Effect of Olive Leaf Extracts on Endothelial Dysfunction in Patients With Acute Coronary Syndrome
Acronym: ACS_ATHEROLIV
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATHEROLIV_ACS
Record Dates: First submitted 2024-11-20; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Acute Coronary Syndrome (ACS); Reactive Hyperemia; Endothelial Dysfunction
Keywords: acute conary syndrome; endothelial dysfunction; olive leaf extract
MeSH Terms: conditions — Acute Coronary Syndrome; Hyperemia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three groups:
  Intervention Group 1:Patients in this group will receive the study drug (olive leaf extract) at a dose of 500 mg (two capsules) twice daily, for a total of 1000 mg per day, for one month.
  Intervention Group 2:Patients in this group will receive the study drug (olive leaf extract) at a dose of 250 mg (one capsule) twice daily, for a total of 500 mg per day, for one month.
  Control Group:Patients in this group will receive a placebo, with one capsule prescribed twice daily, for one month.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A (Active Comparator): Atherolive simple dose
  Interventions: Drug: Atherolive 500mg/day
- Arm B (Active Comparator): Atherolive double dose
  Interventions: Drug: Atherolive 1000/day
- Arm C (Placebo Comparator): Palcebo
  Interventions: Drug: Placbo_Atherolive

INTERVENTIONS:
Drug: Atherolive 500mg/day — Patients will receive a study drug (olive leaf extracts) which will be prescribed at dose of 250 mg (one capsule ) twice daily ( total500mg daily) for one month.
  patients will be assigned to one of three arm using a computer-generated randomization list ( 1:1:1 allocation ).
  Arms: Arm A
Drug: Atherolive 1000/day — Patients will receive a study drug (olive leaf extracts) which will be prescribed at dose of 500 mg (two capsule ) twice daily ( total 1000mg daily) for one month.
  patients will be assigned to one of three arm using a computer-generated randomization list ( 1:1:1 allocation ).
  Arms: Arm B
Drug: Placbo_Atherolive — Patients will receive placebo which will be prescribed one capsule twice daily for one months.
  patients will be assigned to one of three arm using a computer-generated randomization list ( 1:1:1 allocation ).
  Arms: Arm C

SUMMARY:
the study aims to examine the short-term (30 days) effects of olive leaf extract on endothelial function in patients with acute coronary syndrome (ACS).

This investigation will be conducted on patients admitted to the emergency department for ACS. All participants will be screened and included within 24 hours post-ACS event and prior to discharge from the emergency department.

ELIGIBILITY:
Inclusion Criteria:

Age over 18 years. Patients presenting with ST-segment alterations at rest, including ST elevation, with or without troponin elevation.

Patients who have not undergone surgery or have no additional primary percutaneous coronary intervention (P-PCI) planned within 8 weeks from the initial P-PCI.

Patients who provide informed consent. Patients available for and willing to adhere to follow-up procedures. Patients without significant cognitive impairment. Patients with a life expectancy of at least 2 years.

Exclusion Criteria:

* Severe LV hypertrophy (>15 mm);
* Patients with any evidence of inflammatory or malignant disease.
* Patient having valvular heart disease, pacemaker; cardiogenic shock
* Patient having any serious non-cardiac disease associated with a life expectancy <1 year
* Patients undergoing surgery within 30 days
* Patient having gastrointestinal disorder such as Crohn's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) | 30-day
  Change in endothelial function will be evaluated using Reactive Hyperemia Index (RHI) via Peripheral Arterial Tonometry (PAT), measured at baseline and after drug administration (olive leaf extract) in patients with acute coronary syndrome.

SECONDARY OUTCOMES:
MACE rate | 30-day
  -The MACE (Major Adverse Cardiovascular Events) rate will include the following components: Myocardial infarction readmission Nonfatal stroke readmission Cardiovascular death Coronary revascularization, including percutaneous coronary intervention (PCI) and coronary artery bypass grafting (CABG) Admission for heart failure

IPD SHARING:
Plan to Share IPD: No